CLINICAL TRIAL: NCT04670926
Title: Immunosuppression Management in Renal Transplant Recipients With Transplant Excellence Based on TruGraf Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Transplant Genomics, Inc. (Industry)
Collaborators: California Pacific Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: TGRP07
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Kidney Transplant Rejection; Immunosuppression
Keywords: kidney transplant; immunosuppression; biomarkers
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- TruGraf - Group 1: (Experimental): Patients randomized to Group 1 will receive serial TruGraf testing at months 3, 4, 5, 6, 7, 8, 9, and 12. Results will be available in real-time and used by the physician to guide management of immunosuppression.
  Interventions: Diagnostic Test: TruGraf
- CPMC Standard of Care - Group 2: (Active Comparator): Patients randomized to Group 2 or CPMC Standard of Care Group patients will have current standard of care laboratory assessments.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Diagnostic Test: TruGraf — TruGraf results will be available in real-time and used by the physician in conjunction with other standard of care labs to guide management of immunosuppression as follows:
  Patients with a stable serum creatinine and eGFR of > 45 mL/min who also have a TruGraf TX result at month 3 will have their Mycophenolate Mofetil or Mycophenolate Sodium decreased from a standard dose of 1000 mg twice daily to 500 mg twice daily or 720 mg twice daily to 360 mg twice daily respectively.
  Patients with a stable serum creatinine and estimated eGFR of > 45 mL/min who also have a TruGraf TX result at months 4, 5, and 6 will have their Tacrolimus target trough level decreased to a target between 3 and 6.
  Patients with TruGraf not-TX will have no further immunosuppression reduction and continued to be monitored.
  Other Names: TruGraf Blood Gene Expression Test
  Arms: TruGraf - Group 1:
Other: Standard of Care — Patient's immunosuppression will be managed per the current CPMC standard of care that includes continuation of Mycophenolate Mofetil or Mycopheonolate Sodium at 1000 mg bid or 720 mg bid respectively. The dose may be decreased at the discretion of the physician for drug adverse effects such as diarrhea or other gastrointestinal side-effects or neutropenia as is the standard of care. Patients will be maintained on Tacrolimus at target levels that are considered standard of care by the managing physician.
  Arms: CPMC Standard of Care - Group 2:

SUMMARY:
This is an investigator-initiated, single-center, prospective, randomized, proof of concept study. In this study patients who are status post kidney transplantation and meet the inclusion and exclusion criteria will undergo immunosuppression reduction and will be followed closely to assess stability of graft function.

DETAILED DESCRIPTION:
The study will consist of 2 parts (Part-I and Part-II). In Part I of the study, kidney transplant recipients who are low-risk for rejection and meet the inclusion and exclusion criteria for study Part-I will be approached for informed consent in the peri-transplant period, defined as 7 days before to 5 days after transplantation. Basic clinical history and kidney transplant function that are reviewed for routine transplant care are utilized to screen patients who are approached for study discussion and informed consent.

Patients who agree to participation in the study will have received Thymoglobulin induction of at least 4.5 mg/Kg body weight total dose. These patients will have their corticosteroids withdrawn by day 30 post-transplantation and will be followed with kidney function labs at least weekly through day-90 post-transplantation. Withdrawal of corticosteroids in patients who are immunologically at low risk for acute rejection similar to this study population and have received at least 4.5 mg/kg total dose of Thymoglobulin is standard practice. Patients meeting inclusion and exclusion criteria for Part-II of the study will continue with the study. Those failing to meet the inclusion/exclusion criteria for Part-II of the study will conclude the study and will be followed per CPMC standard of care.

In Part II, study patients will be randomized to one of the two groups in a 2:1 ratio. Two patients will be randomized to the study group for every one patient to the standard of care group. A total of 75 patients will be enrolled. Fifty to the study group and 25 to the standard of care group. The patients will have post transplantation follow-up labs as standard of care and clinic visits also as standard of care. There are no additional clinic visits for the study purposes or study procedures. TruGraf blood will be collected at the same time as the standard of care blood tests and additional phlebotomy is not required.

ELIGIBILITY:
Part-I

Inclusion Criteria: Patients who meet all of the following criteria are eligible for enrollment:

1. All males or females of at least 18 years of age.
2. Have the ability to understand the requirements of the study and are able to provide written informed consent.
3. Recipient of a primary deceased-donor or living donor kidney transplant.
4. Patients at low-immunological risk for acute rejection defined as cPRA of less than 50; no DSA; non-African American recipients
5. HLA crossmatch negative (virtual cross match acceptable)
6. Allograft from a deceased donor with KDPI < 50%

Exclusion Criteria: Patients who meet any of the following criteria are not eligible for enrollment:

1. Inability or unwillingness to provide informed consent.
2. Need for combined organ transplantation with an extra-renal organ transplant.
3. Recipients of previous non-renal solid organ and/or islet cell transplantation.
4. Infection with HIV
5. Patients with Hepatitis B or C PCR positive.
6. Patients on corticosteroids at the time of transplantation
7. Patients with leucopenia (WBC <3.0) and thrombocytopenia (platelets <100)
8. Patients who will NOT receive Thymoglobulin induction (>4.5 mg/kg total dose)
9. HLA-identical living related renal transplant recipients

Part-II

Inclusion Criteria: Patients who meet all of the following criteria are eligible for enrollment:

1. Stable serum creatinine level and estimated eGFR of > 45 mL/min at 90 days post-transplantation
2. Kidney transplant patients who are more than 90 days post-transplant.
3. Patients who have received Thymoglobulin induction therapy (> 4.5 mg/kg) and tolerated corticosteroid withdrawal.

Exclusion Criteria: Patients who meet any of these criteria are not eligible for enrollment:

1. Infection with BK viremia with viral loads 10,000 copies/mL.
2. Patients with proteinuria (urine protein >1 gm/gm of creatinine).
3. Patients diagnosed with acute allograft rejection of any grade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-06-03 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Physicians decided to reduce immunosuppression | Baseline to month 12
  Percent or total number of patients who physicians decided could reduce immunosuppression.
Banff pathology | Baseline to month 12
  Banff pathology will be assessed for all study subjects receiving a biopsy during the study period (if performed).
Cost of patient care | Baseline to month 12
  The cost of patient care will be evaluated by measuring the total health care spending for health care services provided during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Ram Peddi, Principal Investigator — California Pacific Medical Center; Patty West-Thielke, PharmD, Study Director — Eurofins-TGI
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rana A, Gruessner A, Agopian VG, Khalpey Z, Riaz IB, Kaplan B, Halazun KJ, Busuttil RW, Gruessner RW. Survival benefit of solid-organ transplant in the United States. JAMA Surg. 2015 Mar 1;150(3):252-9. doi: 10.1001/jamasurg.2014.2038. PMID 25629390
- [Background] Matas AJ, Gillingham KJ, Humar A, Kandaswamy R, Sutherland DE, Payne WD, Dunn TB, Najarian JS. 2202 kidney transplant recipients with 10 years of graft function: what happens next? Am J Transplant. 2008 Nov;8(11):2410-9. doi: 10.1111/j.1600-6143.2008.02414.x. PMID 18925907
- [Background] Lamb KE, Lodhi S, Meier-Kriesche HU. Long-term renal allograft survival in the United States: a critical reappraisal. Am J Transplant. 2011 Mar;11(3):450-62. doi: 10.1111/j.1600-6143.2010.03283.x. Epub 2010 Oct 25. PMID 20973913
- [Background] Montgomery RA. One kidney for life. Am J Transplant. 2014 Jul;14(7):1473-4. doi: 10.1111/ajt.12772. Epub 2014 May 9. No abstract available. PMID 24816339
- [Background] Waldmann H. Drug minimization in transplantation: an opinion. Curr Opin Organ Transplant. 2014 Aug;19(4):331-3. doi: 10.1097/MOT.0000000000000099. No abstract available. PMID 24991978
- [Background] Racusen LC, Solez K, Colvin RB, Bonsib SM, Castro MC, Cavallo T, Croker BP, Demetris AJ, Drachenberg CB, Fogo AB, Furness P, Gaber LW, Gibson IW, Glotz D, Goldberg JC, Grande J, Halloran PF, Hansen HE, Hartley B, Hayry PJ, Hill CM, Hoffman EO, Hunsicker LG, Lindblad AS, Yamaguchi Y, et al. The Banff 97 working classification of renal allograft pathology. Kidney Int. 1999 Feb;55(2):713-23. doi: 10.1046/j.1523-1755.1999.00299.x. PMID 9987096
- [Background] Rush D, Nickerson P, Gough J, McKenna R, Grimm P, Cheang M, Trpkov K, Solez K, Jeffery J. Beneficial effects of treatment of early subclinical rejection: a randomized study. J Am Soc Nephrol. 1998 Nov;9(11):2129-34. doi: 10.1681/ASN.V9112129. PMID 9808101
- [Background] Burghardt KM, Wales PW, de Silva N, Stephens D, Yap J, Grant D, Avitzur Y. Pediatric intestinal transplant listing criteria - a call for a change in the new era of intestinal failure outcomes. Am J Transplant. 2015 Jun;15(6):1674-81. doi: 10.1111/ajt.13147. Epub 2015 Mar 23. PMID 25809131
- [Background] Legendre C, Thervet E, Skhiri H, Mamzer-Bruneel MF, Cantarovich F, Noel LH, Kreis H. Histologic features of chronic allograft nephropathy revealed by protocol biopsies in kidney transplant recipients. Transplantation. 1998 Jun 15;65(11):1506-9. doi: 10.1097/00007890-199806150-00020. PMID 9645814
- [Background] Choi BS, Shin MJ, Shin SJ, Kim YS, Choi YJ, Kim YS, Moon IS, Kim SY, Koh YB, Bang BK, Yang CW. Clinical significance of an early protocol biopsy in living-donor renal transplantation: ten-year experience at a single center. Am J Transplant. 2005 Jun;5(6):1354-60. doi: 10.1111/j.1600-6143.2005.00830.x. PMID 15888041
- [Background] Seron D, Moreso F. Protocol biopsies in renal transplantation: prognostic value of structural monitoring. Kidney Int. 2007 Sep;72(6):690-7. doi: 10.1038/sj.ki.5002396. Epub 2007 Jun 27. PMID 17597702
- [Background] Heilman RL, Devarapalli Y, Chakkera HA, Mekeel KL, Moss AA, Mulligan DC, Mazur MJ, Hamawi K, Williams JW, Reddy KS. Impact of subclinical inflammation on the development of interstitial fibrosis and tubular atrophy in kidney transplant recipients. Am J Transplant. 2010 Mar;10(3):563-70. doi: 10.1111/j.1600-6143.2009.02966.x. Epub 2010 Feb 1. PMID 20121731
- [Background] Rush DN, Henry SF, Jeffery JR, Schroeder TJ, Gough J. Histological findings in early routine biopsies of stable renal allograft recipients. Transplantation. 1994 Jan;57(2):208-11. doi: 10.1097/00007890-199401001-00009. PMID 8310509
- [Background] Kirk AD, Jacobson LM, Heisey DM, Radke NF, Pirsch JD, Sollinger HW. Clinically stable human renal allografts contain histological and RNA-based findings that correlate with deteriorating graft function. Transplantation. 1999 Nov 27;68(10):1578-82. doi: 10.1097/00007890-199911270-00024. PMID 10589958
- [Background] Moreso F, Ibernon M, Goma M, Carrera M, Fulladosa X, Hueso M, Gil-Vernet S, Cruzado JM, Torras J, Grinyo JM, Seron D. Subclinical rejection associated with chronic allograft nephropathy in protocol biopsies as a risk factor for late graft loss. Am J Transplant. 2006 Apr;6(4):747-52. doi: 10.1111/j.1600-6143.2005.01230.x. PMID 16539631
- [Background] Kee TY, Chapman JR, O'Connell PJ, Fung CL, Allen RD, Kable K, Vitalone MJ, Nankivell BJ. Treatment of subclinical rejection diagnosed by protocol biopsy of kidney transplants. Transplantation. 2006 Jul 15;82(1):36-42. doi: 10.1097/01.tp.0000225783.86950.c2. PMID 16861939
- [Background] Lo DJ, Kaplan B, Kirk AD. Biomarkers for kidney transplant rejection. Nat Rev Nephrol. 2014 Apr;10(4):215-25. doi: 10.1038/nrneph.2013.281. Epub 2014 Jan 21. PMID 24445740
- [Background] Kurian SM, Heilman R, Mondala TS, Nakorchevsky A, Hewel JA, Campbell D, Robison EH, Wang L, Lin W, Gaber L, Solez K, Shidban H, Mendez R, Schaffer RL, Fisher JS, Flechner SM, Head SR, Horvath S, Yates JR, Marsh CL, Salomon DR. Biomarkers for early and late stage chronic allograft nephropathy by proteogenomic profiling of peripheral blood. PLoS One. 2009 Jul 10;4(7):e6212. doi: 10.1371/journal.pone.0006212. PMID 19593431
- [Background] Nakorchevsky A, Hewel JA, Kurian SM, Mondala TS, Campbell D, Head SR, Marsh CL, Yates JR 3rd, Salomon DR. Molecular mechanisms of chronic kidney transplant rejection via large-scale proteogenomic analysis of tissue biopsies. J Am Soc Nephrol. 2010 Feb;21(2):362-73. doi: 10.1681/ASN.2009060628. Epub 2010 Jan 21. PMID 20093355
- [Background] Keslar KS, Lin M, Zmijewska AA, Sigdel TK, Tran TQ, Ma L, Bhasin M, Rao P, Ding R, Ikle DN, Mannon RB, Sarwal MM, Strom TB, Reed EF, Heeger PS, Suthanthiran M, Fairchild RL. Multicenter evaluation of a standardized protocol for noninvasive gene expression profiling. Am J Transplant. 2013 Jul;13(7):1891-7. doi: 10.1111/ajt.12284. PMID 23802725
- [Background] Li L, Khatri P, Sigdel TK, Tran T, Ying L, Vitalone MJ, Chen A, Hsieh S, Dai H, Zhang M, Naesens M, Zarkhin V, Sansanwal P, Chen R, Mindrinos M, Xiao W, Benfield M, Ettenger RB, Dharnidharka V, Mathias R, Portale A, McDonald R, Harmon W, Kershaw D, Vehaskari VM, Kamil E, Baluarte HJ, Warady B, Davis R, Butte AJ, Salvatierra O, Sarwal MM. A peripheral blood diagnostic test for acute rejection in renal transplantation. Am J Transplant. 2012 Oct;12(10):2710-8. doi: 10.1111/j.1600-6143.2012.04253.x. PMID 23009139
- [Background] Suthanthiran M, Schwartz JE, Ding R, Abecassis M, Dadhania D, Samstein B, Knechtle SJ, Friedewald J, Becker YT, Sharma VK, Williams NM, Chang CS, Hoang C, Muthukumar T, August P, Keslar KS, Fairchild RL, Hricik DE, Heeger PS, Han L, Liu J, Riggs M, Ikle DN, Bridges ND, Shaked A; Clinical Trials in Organ Transplantation 04 (CTOT-04) Study Investigators. Urinary-cell mRNA profile and acute cellular rejection in kidney allografts. N Engl J Med. 2013 Jul 4;369(1):20-31. doi: 10.1056/NEJMoa1215555. PMID 23822777
- [Background] Kurian SM, Williams AN, Gelbart T, Campbell D, Mondala TS, Head SR, Horvath S, Gaber L, Thompson R, Whisenant T, Lin W, Langfelder P, Robison EH, Schaffer RL, Fisher JS, Friedewald J, Flechner SM, Chan LK, Wiseman AC, Shidban H, Mendez R, Heilman R, Abecassis MM, Marsh CL, Salomon DR. Molecular classifiers for acute kidney transplant rejection in peripheral blood by whole genome gene expression profiling. Am J Transplant. 2014 May;14(5):1164-72. doi: 10.1111/ajt.12671. Epub 2014 Apr 11. PMID 24725967
- [Background] Haas M, Sis B, Racusen LC, Solez K, Glotz D, Colvin RB, Castro MC, David DS, David-Neto E, Bagnasco SM, Cendales LC, Cornell LD, Demetris AJ, Drachenberg CB, Farver CF, Farris AB 3rd, Gibson IW, Kraus E, Liapis H, Loupy A, Nickeleit V, Randhawa P, Rodriguez ER, Rush D, Smith RN, Tan CD, Wallace WD, Mengel M; Banff meeting report writing committee. Banff 2013 meeting report: inclusion of c4d-negative antibody-mediated rejection and antibody-associated arterial lesions. Am J Transplant. 2014 Feb;14(2):272-83. doi: 10.1111/ajt.12590. PMID 24472190